CLINICAL TRIAL: NCT03542513
Title: Detection of Biomarkers in First-void Urine Samples for Follow-up of Women Treated for High-grade Cervical Intraepithelial Neoplasia (CIN)
Brief Title: First-void Urine Samples for the Follow-up of Women Treated for High-grade Cervical Intraepithelial Neoplasia (CIN)
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Pierre Van Damme, Principal Investigator, Universiteit Antwerpen
Other Study IDs: B300201732818
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Cervical Cancer
Keywords: Human Papillomavirus; Biomarker; Self-sampling; First-void urine; Cervical Intraepithelial Neoplasia; LLETZ
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — First-void urine samples, self collected vaginal swabs and physician collected cervical brush samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Colli-Pee — Urine samples will be collected with the Colli-Pee device (Novosanis NV, Wijnegem, Belgium).
Device: Qvintip — Vaginal self-samples will be collected with the Qvintip (Aprovix AB, Uppsala, Sweden).

SUMMARY:
The aim of this study is to analyse biomarkers in first-void urine for improved follow-up of women treated for high grade cervical intraepithelial neoplasia (CIN).

DETAILED DESCRIPTION:
In total 100 women, diagnosed with CIN2/3 and scheduled for LLETZ (Large Loop Excision of the Transformation Zone), will be included in this trial. These women are asked to collect two FV urine samples with the Colli-Pee device (Novosanis, Wijnegem, Belgium) prior to their treatment (one at home and one at the hospital) and at five additional time points post treatment (1-3-6-12-24 months) at home. In addition, five self-collected vaginal swabs will be taken, two before treatment (1 at home and 1 at the hospital) and three (6-12-24 months) after treatment at home. Qvintip devices are used for vaginal self-sampling.

During follow-up visits cervical samples and optional biopsies are collected by the physician and respectively send to the UZA anatomic pathology unit to determine the patient's HPV status, cytology and histology. For the study, one extra cervical sample will be taken by the physician just before treatment, that is not part of the normal standard procedure.

ELIGIBILITY:
Inclusion Criteria:

* Female (18 years and older)
* Scheduled for LLETZ treatment of diagnosed, histologically confirmed high grade CIN lesions
* Giving informed consent to the research team (CEV) to contact his/her GP and/or gynaecologist to access details of the participants HPV vaccination (schedule) and results of cervical smears/cytology, HPV tests, colposcopy, and biopsy.
* Not participating in another clinical study where a drug or biological is administered.
* Able to understand the information brochure/what the study is about.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The cohort involves 100 women, diagnosed with histologically confirmed high grade CIN lesions requested for LLETZ treatment. Before this treatment an extra cervical sample is collected by the clinician. In addition, these women are asked to collect first-void urine samples with the Colli-Pee device, vaginal samples with the Qvintip device and to fill in a questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
hrHPV DNA status of self-collected first-void urine and vaginal samples vs physician sampled cervical specimens. | Within 6 months after study completion
  Concordance hrHPV DNA status of self-collected first-void urine and vaginal samples from women treated for high-grade cervical lesions to that of physician sampled cervical specimens.

SECONDARY OUTCOMES:
hrHPV DNA status of self-collected first-void urine and vaginal samples at home vs at the hospital. | Within 6 months after study completion
  Concordance hrHPV DNA status of self-collected first-void urine and vaginal fluid samples at home to self-collected samples at the hospital.
Effect of treatment on HPV DNA presence. | Within 6 months after study completion
  Evaluate the effect of treatment on HPV DNA presence by the use of self-collected first-void urine and vaginal self-sampling for HPV DNA detection.
Validate the performance of additional biomarkers. | Within 6 months after study completion
  Validate the performance of additional biomarkers (mRNA, genotyping, DNA methylation markers, viral load) for further staging of hrHPV infections.
Preference of women for self-sampling methods. | Within 6 months after study completion
  Gather information about the preference of women for first-void urine sample collection compared vaginal self-sampling methods, and a clinician collected sample (smear).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, Principal Investigator — Centre for the Evaluation of Vaccination
Locations (1):
- University of Antwerp - Centre for the Evaluation of Vaccination, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No